CLINICAL TRIAL: NCT05989386
Title: Outcomes of High-volume Saline Irrigation VS Povidone-Iodine Solution Cleaning of Intraoperative Incision Wound in Preventing Surgical Site Infections in Emergency Laparotomies: A Randomized Controlled Trial
Brief Title: Outcomes of High-volume Saline Irrigation VS Povidone-Iodine Solution Cleaning of IOWI in Preventing SSIs in Emergency Laparotomies
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Omer bin khalid, Principal Investigator (Assistant Professor), Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2811
Record Dates: First submitted 2023-07-19; First posted 2023-08-14 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Surgical Site Infection; Surgical Wound; Surgical Incision; Emergency Laparotomies; Laparotomies; Post Operative Wound Infection; Wound Infection; Seroma
MeSH Terms: conditions — Surgical Wound Infection; Surgical Wound; Wound Infection; Seroma | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Intra-operative wound irrigation of 0.9% solution saline solution
  Interventions: Procedure: 0.9% saline solution
- Group B (Active Comparator): No intra-operative wound lavage done
  Interventions: Procedure: Povidone-iodine Swab

INTERVENTIONS:
Procedure: 0.9% saline solution — During emergency laparotomy, after the primary surgical procedure. the sheath will be sutured and the incision site will then be irrigated with three rounds of 1 liter of 0.9% saline solution, which will be completely aspirated before the closure of the incisional wound in experimental group.
  Arms: Group A
Procedure: Povidone-iodine Swab — No intra-operative wound lavage done, and wound would be cleaned with povidone doused swab.
  Other Names: Control
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to compare the outcomes of High-volume saline irrigation vs Povidone-iodine solution cleaning of the intraoperative incision wound in preventing superficial surgical site infections in patients undergoing emergency laparotomies. The main question it aims to answer are:

* Incidence of SSI after intervention
* Length of hospital stay

Participants will be randomly assigned to two groups receiving either of the two groups:

Group A: 1000ml of IOWI with saline solution prior to incision closure Group B: The incisional wound will be closed conventionally without irrigation.

Researchers will compare groups A( experimental group) and B (control group) to compare the incidence of superficial surgical site infections after intervention.

ELIGIBILITY:
Inclusion Criteria:

* • Patients undergoing emergency laparotomy under the care of surgical-6 unit of Dr. Ruth K. M. Pfau Civil Hospital Karachi

  * The age of patients should be between 18-60 years old.

Exclusion Criteria:

* Diabetic patients
* Immune-suppressed patients
* Patients taking steroids
* Patients undergoing chemo-radiotherapy.
* Pregnant females
* Previous abdominal surgery within the last 30 days.
* Presence of concurrent abdominal wall infections.
* Trauma Laparotomies
* Large Bowel perforations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Superficial Surgical site infections | Upto 4 weeks post-operatively
  Development of Superficial Surgical Site Infection as determined by the CDC guidelines.

SECONDARY OUTCOMES:
Length of Hospital Stay | Upto 4 weeks post-operatively
  Number of in-hospital days (from time of admission to time of discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bin Khalid, Assist Prof., Principal Investigator — Dr. Ruth F. M. Pfau Civil Hospital Karachi; Imrana Zulfikar, Professor, Study Director — Dr. Ruth F. M. Pfau Civil Hospital Karachi
Locations (1):
- Dr. Ruth K. M. Pfau Civil Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No